CLINICAL TRIAL: NCT04478201
Title: Comparing the Effectiveness of Side-lying Sleep Positioning to Back-lying at Reducing Oxygen Desaturation Resulting From Obstructive Sleep Apnoea in Infants With Cleft Palate
Brief Title: Comparing the Side-lying Sleep Positioning to Back-lying in Infants With Cleft Palate
Acronym: SLUMBRS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other); Centre for Trials Research, Cardiff University (Unknown); University College, London (Other); Cleft Lip and Palate Association (Unknown); University Hospital Southampton NHS Foundation Trust (Other); Salisbury NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B00785
Record Dates: First submitted 2020-05-28; First posted 2020-07-20 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Obstructive Sleep Apnea; Cleft Palate
Keywords: Sleep; Sleep position; Infants with cleft palate
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cleft Palate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back lying sleep position (Experimental): sleep on the back
  Interventions: Other: back sleep positioning
- Side lying sleep position (Experimental): sleep on the side
  Interventions: Other: side sleep positioning

INTERVENTIONS:
Other: back sleep positioning — sleeping on the back.
  Arms: Back lying sleep position
Other: side sleep positioning — sleeping on the side
  Arms: Side lying sleep position

SUMMARY:
The craniofacial abnormalities found in infants and children with cleft palate (CP) lead to increased risk of obstructive sleep apnoea (OSA). In children and adults sleep position is known to influence the patency of the airway during sleep. Altering sleep position in infants with CP may offer a 'low-cost, high impact' intervention to limit the negative impacts of OSA on child development.

Children with CP are at increased risk of impairment in learning, memory and cognition, with OSA representing an additional risk to cognitive development. Infants with CP are at risk of poor weight gain and 'failure to thrive', which can be further exacerbated by co-existing OSA.

The design and conduct of the proposed randomised controlled trial will benefit from lessons learned from both the feasibility and other previous studies. Investigators demonstrated that existing advice given about sleep position varied significantly with some centres recommending back-lying and others side-lying. Sample size calculations were based on this multi-source data. Parents in the feasibility study knew that sleep position advice for infants with CP changes regularly. They understood why not adhering to 'national guidance' (DoH 2009, Back to Sleep) could be necessary as their infants are "different to normal infants".

How will this study benefit infants with cleft palate and their parents? The proposed study will eliminate the current uncertainty and variability in advice provided to parents of infants with CP, whilst potentially limiting the negative impact of OSA on development. This work has been prioritised and received unanimous support from Cleft Lip and Palate Association (CLAPA), Craniofacial Society Great Britain and Ireland (CFSGBI) and Clinical Nurse Specialists. Aim.To determine the clinical effectiveness in infants with CP of side-lying as compared to back-lying sleep positioning in reducing oxygen desaturation resulting from OSA.

DETAILED DESCRIPTION:
The primary aim of this project is to determine the clinical effectiveness in infants with cleft palate (CP) of side-lying as compared to back-lying sleep positioning in reducing oxygen desaturation resulting from obstructive sleep apnoea (OSA). This will be achieved:

* comparing oxygen saturation during sleep in the side- and back-lying positions at 1 month of age.
* comparing sleep quality between the side-lying and back-lying groups using a parental questionnaire.
* co-developing national recommendations with parents regarding sleep position for infants with CP.

A randomised controlled trial (RCT) of side-lying compared with back-lying sleep positioning in reducing oxygen desaturation resulting from OSA in infants with CP. The design and conduct of the study will benefit from lessons learned from the feasibility and other previous studies. All parents in the feasibility study indicated strong interest to participate in further studies evaluating the effects of sleep position. Infants meeting the eligibility criteria will be randomised to side-lying or back-lying in a ratio 1:1 using a minimisation routine incorporating a random element to reduce predictability. Minimisation factors will be clinical site and syndrome suspected or indicated (yes / no). Allocations will be delivered via a password-protected web-based system. The allocated position will only be used on the day(s) when the infant is monitored for the study purposes. Thereafter, parents will be free to revert back to the standard sleep position as advised by their cleft centre, should it be different than that used for the monitoring period. All centres represented at the preparatory meeting with the United Kingdom (UK) Lead Clinical Nurse Specialist group, confirmed that the side-lying position was recommended in some infants at their centre, irrespective of whether it was the standard advice used. As such, all centres had experience of the side-lying position. It was decided not to change the specific advice that centres give to parents regarding how to position the infant in a side-lying position, but any standard written or verbal information would be collected by the study documents.

An internal pilot will investigate participants' opinions about their participation in the study. Using bespoke questionnaires participants' experience will be assessed and it will be decided how it could be improved. After 6 months questionnaire results will be analysed and if necessary study amendments will be put in place to reflect participants' opinions.

Data from the feasibility study and published studies have reported estimates of the standard deviation (SD) of the primary outcome ODI-4 in the side-lying infants at four weeks to range from 8 to 11 units, with a higher SD observed in the back-lying group. The observed difference in mean ODI-4 between the side-lying and back-lying infant cohorts was 15 units (a standardised effect size of 0.91). Investigators considered a smaller but more realistic difference in means of five units to be a clinically important difference (SD 10), a standardised effect size of 0.5. The sample size calculation comparing two means with unequal variances for the primary outcome was, therefore, based on a standardised effect size of 0.5. To account for potential unequal variances in each group a variance ratio of 2 was used in the calculations. To detect a difference of 0.5 standard deviation score (SDS) with 80% power and alpha equal to 0.05 would require 96 infants to be monitored in each arm of the trial (a total of 192 participants). Informed by the multicentre feasibility and oximetry studies the sample size will be inflated to 244 participants in the RCT, to allow for potential attrition of 21%.

This will follow a pre-specified and approved statistical analysis plan. The primary analysis of the RCT data will use intention-to-treat. Baseline data will be analysed to assess the comparability of the demographic and clinical characteristics of the participants. Data from the trial arms will be compared using generalised linear models and adjusted for minimisation covariates where appropriate. Estimates of treatment effect size will be reported as differences in means for continuous outcomes, and risk ratios for dichotomous outcomes and reported along with 95% confidence intervals. Subgroup analyses will explore the effects of sleep position on infants with and without suspected associated syndromes through subgroup treatment interactions, at a stricter alpha level 0.01.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with an isolated CP under the care of a collaborating centre
* Infants who are 3 to 5 weeks of age when monitored
* Parents willing to give consent and able to complete study procedures

Exclusion Criteria:

* Infants with associated cleft lip
* Infants born prematurely (before 37 week gestation or up to and including 36 weeks and 6 days)
* Infants with cardiorespiratory disease
* Infants requiring an intervention to assist with breathing (nasopharyngeal airway)
* Infants requiring an intervention to assist with feeding (nasogastric tube)

Ages: 21 Days to 35 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation during sleep at 1 month of age | 1 month of age
  Oxygen saturation during sleep at 1 month of age (expressed as 4% oxygen desaturation index, ODI-4). Oximetry is considered the mainstay of assessment of oxygenation in infants and will be the primary outcome measurement instrument. The ODI-4 represents the average number of times that oxygen saturation falls by at least 4% from baseline every hour.

SECONDARY OUTCOMES:
SPO2 mean | completed at 1 month
  mean oxygen saturation
SPO2 nadir | completed at 1 month
  nadir oxygen saturation
Total sleep time | completed at 1 month.
  the proportion of total sleep time (TST) with oxygen saturation below: 97%, 95%, 90% and 80%
Oxygen saturation during sleep at 1 month of age | 1 month of age
  Oxygen saturation during sleep at 1 month of age (expressed as 3% oxygen desaturation index, ODI-3). Oximetry is considered the mainstay of assessment of oxygenation in infants and will be the primary outcome measurement instrument. The ODI-3 represents the average number of times that oxygen saturation falls by at least 3% from baseline every hour.
Weight | completed at 1 month.
  child's weight
Length | 1 month of age
  participant's length
Head circumference | 1 month of age
  participant's head circumference
Number of participants with Adverse events. | From consent for up to 2 weeks
  Number of participants experiencing Adverse events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Iain Bruce, Prof, Study Director — Manchester University NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Birmingham Women'S and Children'S Nhs Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children'S Nhs Foundation Trust, Liverpool
  - Great Ormond Street Hospital For Children Nhs Foundation Trust, London
  - Manchester University Nhs Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Salisbury Nhs Foundation Trust, Salisbury
  - Swansea Bay University Local Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metryka A, Cuniffe C, Evans HJ, Gavlak JG, Hudson N, Kirby N, Lakhanpaul M, Lin YL, Murray C, Rajai A, Robson H, Schilder A, Walsh T, Bruce I. Study protocol for randomised clinical trial comparing the effectiveness of side-lying sleep positioning to back-lying at reducing oxygen desaturation resulting from obstructive sleep apnoea in infants with cleft palate (SLUMBRS2). BMJ Open. 2021 Apr 7;11(4):e049290. doi: 10.1136/bmjopen-2021-049290. PMID 33827851